CLINICAL TRIAL: NCT04925297
Title: The Characteristics of Neurological Sequelae in Patients With Acute Carbon Monoxide Poisoning
Brief Title: Neurological Sequelae in Patients With Acute Carbon Monoxide Poisoning
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: AF-IRB-030-06
Record Dates: First submitted 2021-05-26; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Carbon Monoxide Poisoning
Keywords: carbon monoxide poisoning; neurological sequelae
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-NS ( Non-neurological sequelae) group: Patients who do not develop neurological dysfunction after acute carbon monoxide poisoning
  Interventions: Other: No intervention
- NS (Neurological sequelae) group: Patients who develop neurological dysfunction after acute carbon monoxide poisoning
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be given

SUMMARY:
The purpose of this study is to access the clinical characteristics and risk factors for neurological sequelae after acute carbon monoxide poisoning.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients meet the inclusion criteria would be given informed consent and entry the study. The data will be collected according to self-designed questionnaire, including :1) The baseline characteristics: would be recorded 6 hours after patients presentation;2) Patients' self evaluation for discomfort symptoms: would be recorded at day 0, week 1, 3 and 6, month 6 and 12；3) Neurological function: would be recorded at day 0, week 6, month 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* patients present within 12 hours after acute carbon monoxide poisoning;
* age older than 16 years.

Exclusion Criteria:

* pregnant women；
* patients receive oxygen therapy before presentation;
* have history of acute carbon monoxide poisoning within 1 year;
* have been diagnosed any of the following disease: Parkinson disease; cognitive disorder, psychiatric disorders, sequelae of cerebral infarction or hemorrhage, chronic kidney disease and receive hemodialysis, congestive heart failure ( NYHA class III-IV)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with acute carbon monoxide poisoning would be recruited from the First Hospital of Jilin University.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Mini-mental State Examination (MMSE) score at 6 weeks | Changes of score from baseline to 6 weeks
  Score ranges from 0 to 30, a lower score means a worse outcome.
Changes of Mini-mental State Examination (MMSE) score at 6 months | Changes of score from baseline to 6 months
  Score ranges from 0 to 30, a lower score means a worse outcome.
Changes of Mini-mental State Examination (MMSE) score at 12 months | Changes of score from baseline to 12 months
  Score ranges from 0 to 30, a lower score means a worse outcome.
Changes of Montreal cognitive assessment (MoCA）score at 6 weeks | Changes of score from baseline to 6 weeks
  Score ranges from 0 to 30, a lower score means a worse outcome.
Changes of Montreal cognitive assessment (MoCA）score at 6 months | Changes of score from baseline to 6 months
  Score ranges from 0 to 30, a lower score means a worse outcome.
Changes of Montreal cognitive assessment (MoCA）score at 12 months | Changes of score from baseline to 12 months
  Score ranges from 0 to 30, a lower score means a worse outcome.
Changes of Hamilton Depression Scale(HAMD) score at 6 weeks | Changes of score from baseline to 6 weeks
  Score ranges from 0 to 54, a higher score means a worse outcome.
Changes of Hamilton Depression Scale(HAMD) score at 6 months | Changes of score from baseline to 6 months
  Score ranges from 0 to 54, a higher score means a worse outcome.
Changes of Hamilton Depression Scale(HAMD) score at 12 months | Changes of score from baseline to 12 months
  Score ranges from 0 to 54, a higher score means a worse outcome.
Changes of Hamilton Anxiety Scale (HAMA) score at 6 weeks | Changes of score from baseline to 6 weeks
  Score ranges from 0 to 56, a higher score means a worse outcome.
Changes of Hamilton Anxiety Scale (HAMA) score at 6 months | Changes of score from baseline to 6 months
  Score ranges from 0 to 56, a higher score means a worse outcome.
Changes of Hamilton Anxiety Scale (HAMA) score at 12 months | Changes of score from baseline to 12 months
  Score ranges from 0 to 56, a higher score means a worse outcome.
Changes of Activity of Daily Living (ADL) score at 6 weeks | Changes of score from baseline to 6 weeks
  Score ranges from 0 to 80, a higher score means a worse outcome.
Changes of Activity of Daily Living (ADL) score at 6 months | Changes of score from baseline to 6 months
  Score ranges from 0 to 80, a higher score means a worse outcome.
Changes of Activity of Daily Living (ADL) score at 12 months | Changes of score from baseline to 12 months
  Score ranges from 0 to 80, a higher score means a worse outcome.
Changes of self-evaluation of discomfort symptoms scale at 1 week | Changes of score from baseline to 1 week
  This is a self designed questionnaire, score ranges from 0 to 66, a higher score means a worse outcome
Changes of self-evaluation of discomfort symptoms scale at 3 weeks | Changes of score from baseline to 3 weeks
  This is a self designed questionnaire, score ranges from 0 to 66, a higher score means a worse outcome
Changes of self-evaluation of discomfort symptoms scale at 6 weeks | Changes of score from baseline to 6 weeks
  This is a self designed questionnaire, score ranges from 0 to 66, a higher score means a worse outcome
Changes of self-evaluation of discomfort symptoms scale at 6 months | Changes of score from baseline to 6 months
  This is a self designed questionnaire, score ranges from 0 to 66, a higher score means a worse outcome
Changes of self-evaluation of discomfort symptoms scale at 12 months | Changes of score from baseline to 12 months
  This is a self designed questionnaire, score ranges from 0 to 66, a higher score means a worse outcome

SECONDARY OUTCOMES:
Rates of cardiovascular and cerebrovascular events | through study completion, an average of 1 year
  Cardiovascular and cerebrovascular events includes：cardiac arrest, myocardial infarction, cerebral hemorrhage, and cerebral infarction. A patient develops any of the former diseases during following up would be record as 1 event.
Rates of accidental injury | through study completion, an average of 1 year
  Accidental injuries may include accidental fall, fracture, traffic accident etc. A patient develops any of the former during following up would be record as 1 event.

CONTACTS AND LOCATIONS:
Overall Officials: Li Pang, M.D., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided
The IPD would be shared with other researcher through e-mail contact with Ning Dong (dnjl2007@jlu.edu.cn)